CLINICAL TRIAL: NCT05328024
Title: Identification of Predictive Factors for the Response to Anti-Programmed Cell Death Protein 1 (PD1) Immunotherapy in Head and Neck Squamous Cell Carcinoma
Acronym: IPRICE
Status: Recruiting | Type: Observational
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: Centre National de la Recherche Scientifique, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-003
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Immunotherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor and blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recurrent and/or metastatic head and neck carcinoma: Patients with indication of anti-PD1 immunotherapy according to recommendations
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Drug: Immunotherapy — anti-PD1

SUMMARY:
This project aims to organise the sampling of blood and tumor at key points of the standard of care of patients with recurrent or metastatic squamous-cell carcinoma of the head and neck (HNSCC). This will allow to identify new potential predictive biomarkers of efficacy of immunotherapy and to investigate the evolution of the tumoral microenvironment after successive systemic treatments.

DETAILED DESCRIPTION:
Tumor and blood samples will be collected on patients treated by anti-PD1 immunotherapy at different timepoints. Tumor samples will be collected (i) before initiation of immunotherapy, (ii) at 50 days after initiation of immunotherapy and, optionally, in case of disease progression, (iii) before the initiation of the new line of chemotherapy and (iv) at 50 days after initiation of chemotherapy. Blood samples will be collected : (i) before initiation of immunotherapy, (ii) at each cycles of treatment until 84 days after initiation of immunotherapy and, optionally, in case of disease progression, (iii) before the initiation of the new line of chemotherapy and (iv) at each cycle until 50 days after initiation of chemotherapy (maximum 2 samples per month).

ELIGIBILITY:
Inclusion Criteria:

* Patients with recurrent squamous-cell carcinoma of the head and neck not amenable to local therapy and/or with metastatic disease
* Tumor directly accessible to clinical examination (tumor of oral cavity and of oropharynx) and/or cervical lymphadenopathy accessible to echography allowing to realise biopsy under local anesthesia
* Indication to treatment by anti-PD1 immunotherapy according to French competent authority recommendations
* Performance status 0, 1 or 2
* At least one measurable lesion on RECIST V1.1 criteria

Exclusion Criteria:

* Head and neck squamous cell carcinoma accessible to a local treatment
* Cancer of nasopharynx, sinus or nasal cavity
* Other histology than epidermoid
* Patients with contraindication for anti-PD1 immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with recurrent or metastatic squamous-cell carcinoma of the head and neck not amenable to local therapy and/or with metastatic disease and with an indication to treatment by anti-PD1 immunotherapy
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2029-08-25 (Estimated); Study Completion 2029-08-25 (Estimated)

PRIMARY OUTCOMES:
prospective validation of the expression of interferon-gamma signature to predict anti-PD1 immunotherapy response. | at 3 months after initiation of immunotherapy
  objective response according to RECIST v1.1 (response evaluation criteria in solid tumours)
prospective validation of the expression of interferon-gamma signature to predict anti-PD1 immunotherapy response. | at 3 months after initiation of immunotherapy
  objective response according to iRECIST criteria (immune response evaluation criteria in solid tumours)

SECONDARY OUTCOMES:
Prospective validation of the expression of interferon-gamma signature to predict progression free survival. | at 3 years after inclusion
  Time from date of inclusion to the event of tumor recurrence or clinical progression or radiological progression on primary tumor or on lymph nodes or on metastasis or death whatever the cause.
Prospective validation of the expression of interferon-gamma signature to predict overall survival. | at 3 years after inclusion
  Time from date of inclusion to death whatever the cause.
Prospective validation of the expression of interferon-gamma signature to predict duration of objective response. | at 3 years after inclusion
  Time from date of first observation of objective response to progressive disease according to RECIST v1.1 or death..
Exploratory outcome : investigation of the expression of other molecular signatures such as immune cells panel within the tumor microenvironment to predict anti-PD1 immunotherapy response. | at 3 months after initiation of immunotherapy
  objective response according to RECIST v1.1
Exploratory outcome : investigation of the expression of other molecular signatures such as immune checkpoints protein expression level to predict anti-PD1 immunotherapy response. | at 3 months after initiation of immunotherapy
  objective response according to RECIST v1.1
Exploratory outcome : investigation of the expression of other molecular signatures such as biomarkers expression level involved in immunogenic cell death and in mitophagy to predict anti-PD1 immunotherapy response. | at 3 months after initiation of immunotherapy
  objective response according to RECIST v1.1
Exploratory outcome : investigation of the expression of other molecular signatures such as protein expression level involved in hypoxia to predict anti-PD1 immunotherapy response. | at 3 months after initiation of immunotherapy
  objective response according to RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de cancérologie Strasbourg Europe, Strasbourg, France

REFERENCES:
- [Derived] Helene C, Conrad O, Pflumio C, Borel C, Voegelin M, Bernard A, Schultz P, Onea MA, Jung A, Martin S, Burgy M. Dynamic profiling of immune microenvironment during anti-PD-1 immunotherapy for head and neck squamous cell carcinoma: the IPRICE study. BMC Cancer. 2023 Dec 8;23(1):1209. doi: 10.1186/s12885-023-11672-x. PMID 38066522